CLINICAL TRIAL: NCT06291103
Title: Screening for Subclinical Antibody Mediated Rejection and Efficacy of Belatacept in the Context of de Novo Donor Specific Antibody After Kidney Transplantation (BELA-M-R)
Acronym: BELA-M-R
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/0342/HP
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Kidney Transplant Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): - Experimental arm: conversion to Belatacept CNI will be tapered within 3 months: 75 % of initial dose on the first month, 50 % on the second month, 25 % on the third month, and stopped and a conversion to Belatacept will be performed. It will be administered (6mg/kg) every 2W for the first 2 months and then every month until kidney graft survival.
  Interventions: Drug: Conversion to Belatacep
- Control (Active Comparator): - Control arm: Standard of care treatment (SOC regimen) with Tacrolimus Tacrolimus will be continued until kidney graft survival with objective of whole blood through levels between 6 and 8 ng/mL
  Interventions: Drug: Standard of care treatment (SOC regimen) with Tacrolimus

INTERVENTIONS:
Drug: Conversion to Belatacep — CNI will be tapered within 3 months: 75 % of initial dose on the first month, 50 % on the second month, 25 % on the third month, and stopped and a conversion to Belatacept will be performed. It will be administered (6mg/kg) every 2W for the first 2 months and then every month until kidney graft survival.
  Arms: Experimental
Drug: Standard of care treatment (SOC regimen) with Tacrolimus — Tacrolimus will be continued until kidney graft survival with objective of whole blood through levels between 6 and 8 ng/mL
  Arms: Control

SUMMARY:
Antibody mediated rejection (ABMR) is a major cause of graft loss after kidney transplantation (KT) and is mainly associated with preformed anti-HLA donor specific antibodies (DSAs) (phenotype 1) or de novo DSAs (dnDSAs) (phenotype 2). Preexisting DSA-associated ABMR have superior graft survival compared with dnDSA-associated ABMR, which could partly be explained by the fact that patients with de novo DSA-associated ABMR have biopsy later, when graft dysfunction and/or proteinuria are already present. ABMR is a progressive process with an early stage called subclinical ABMR (sABMR), in which histological lesions are present in the kidney graft without clinical graft dysfunction. These early lesions are now well recognized as risk factors for transplant glomerulopathy and poor graft survival in phenotype 1 ABMR (ref 5). The impact of sABMR associated with dnDSA at any time post-transplant has been less studied and reported. Recently, we published a retrospective multicenter study within the Spiesser Group that included 123 patients without graft dysfunction who underwent graft biopsy because of the presence of dnDSA (One Lambda, MFI > 1000). Performing a kidney graft biopsy after dnDSA indentification without renal dysfunction leads to the diagnosis of active sABMR in 35 % of cases. Nevertheless, we did not observe any effect of standard of care treatment in active sABMR. Very recently, an expert consensus for the recommended treatment for ABMR after KT was published. They concluded the clear lack of evidence but a standard of care for ABMR was nevertheless defined. Therefore, we propose to evaluate a new strategy for active sABMR, testing a conversion from calcineurin inhibitor (CNI) to belatacept associated with the recently recommended standard of care (SOC) compared to continuing CNI. Belatacept might help to manage nonadherence, decrease the toxicity of CNI on an endothelium already affected by microvascular inflammation, and reduce DSA titers.

The monitoring of dnDSA after KT and an indication graft biopsy in case of appearance, even in the absence of graft dysfunction, is not part of a routine clinical practice in all KT centers. This strategy could be a valuable option, in order to begin treatment of ABMR before graft dysfunction occurs, and therefore to improve prognosis associated with phenotype 2 ABMR. Parajuli et al.4 suggested that early diagnosis and treatment of sABMR with SOC, using DSA monitoring may improve outcomes after KT, but this is a retrospective and no-randomized study. This study will be the first prospective randomized study in the context of de novo DSA. We will evaluate a new combination of treatment for ABMR in the context of dnDSA with subclinical lesions and in the same time may help to determine the real incidence of sABMR in KT recipients with subclinical dnDSA. The use of belatacept in the context of sABMR to improve the non-adherence and to decrease the endothelial toxicity had never been evaluated in a prospective way.

ELIGIBILITY:
Inclusion Criteria:

1. Screening inclusion criteria:

   * Kidney transplant recipient
   * Adult
   * De novo DSA (MFI > 1000 using the Luminex single antigen beads assay or positive with the manufacturer criteria according to the Luminex assay) absent on the day of kidney transplantation and in the sera prior to kidney transplantation
   * No clinical graft dysfunction at time of DSA detection (< 20 % variation of eGFR compared to last 3 months before detection and < 0,5 g/g proteinuria/creatinuria ratio)
   * Affiliation with, or beneficiary of a Social security (national health insurance) category
   * Person having read and understood the information letter and signed the consent form
   * Women of childbearing potential with effective contraception/very-effective contraception (Cf. CTFG) (oestro-progestatives or intra-uterine device or tubal ligation) and a negative blood pregnancy test.
   * Women surgically sterile (absence of ovaries and/or uterus)
   * Postmenopausal women: confirmation diagnostic (non-medically induced amenorrhea for at least 12 months prior to the inclusion visit)
2. Randomization inclusion criteria:

   * Patients with active sABMR, according Banff 2019 classification, with very slight transplant glomerulogathy (cg = 0 or 1).

Exclusion Criteria:

1. Screening exclusion criteria:

   * Minor
   * Specific treatment for DSA occurrence before kidney graft biopsy: IVIG or rituximab or plasmapheresis or immunoabsorption
   * ABO incompatible kidney transplantation
   * Combined transplantation
   * Transplant recipients who are Epstein-Barr virus (EBV) seronegative or serostatus unknown.
   * Hypersensitivity to the active substance or to any of the excipients - Pregnant or parturient or breastfeeding woman or absence of contraception
   * Person deprived of liberty by an administrative or judiciary decision or person placed under judicial protection, under guardianship or supervision
   * Person consenting to the research participating to another trial
   * Medical history or psychological or sensorial abnormality prone to inhibit the subject to understand the conditions required for his/her participation to the protocol or unable him/her to give an informed consent
   * No signed ICF
2. Randomization exclusion criteria:

   * No sABMR or chronic active sABMR (cg > 1) on initial biopsy
   * History of severe opportunistic infection before randomization
   * Acute or chronic infection with HBV, HCV or HIV
   * EBV negative serology
   * History of post-transplant lymphoproliferative disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2031-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
The efficacy of belatacept combined with standard of care, compared to calcineurin inhibitors (CNI) combined with standard of care, among kidney transplant recipients with sABMR | over 12 months post-biopsy
  Proportion in each arm, at 12 months post randomization, of patients with:
  * decrease eGFR > 20% at 12 months post randomization, according to CKD-EPI formula
  * or bad features on 12-month protocol biopsy: cg > 1
  * or chronic active ABMR according Banff 2019 classification,
  * or < 50 % MFI reduction of DSA,
  * or proteinuria/creatinuria ratio > 0.5 g/g,
  * or death,
  * or graft loss.